CLINICAL TRIAL: NCT00344084
Title: Active Surveillance for Cutaneous Leishmaniasis in Mali
Brief Title: Surveillance for Leishmaniasis Skin Lesions in Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906121; 06-I-N121
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2012-09-17

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Leishmania Major; Phlebotomus Duboscqi; Dermatology; Vector-Transmitted Disease; Africa; Cutaneous Leishmaniasis; CL
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Vector Borne Diseases

SUMMARY:
This study will examine why some people who become infected with the leishmaniasis parasite develop skin lesions and others do not. The parasite that causes leishmaniasis is transmitted by the bite of a sandfly. It can cause skin lesions that may persist for several months, spread to other parts of the body, and become infected with bacteria. Treated with medicine, leishmaniasis can be cured completely.

People 1 year of age and older who live in the Mali villages of Kemena or Sougoula may be eligible for this study.

Participants are injected with a small amount of inactive parasites into the skin of their arm. People who have a reaction to the test, and thus have been exposed to the parasite, are examined for skin lesions. Their lesions, if any, are evaluated and treated, and their participation in the study ends.

Participants who do not react to the skin test are examined for skin lesions every month for 5 months. Those who are 18 years of age or older and have mild leishmaniasis skin lesions may have a small amount of fluid injected into a lesion in order to remove parasites for laboratory analysis.

Patients' lesions may be photographed to compare what they look like before and after treatment. Lesions are treated with an ointment containing an antibiotic and a disinfectant twice a day for 20 days. The lesions are examined 1 and 3 weeks after treatment is completed to see if the disease has been cured. A few months later, the skin test is repeated to determine whether the person has been exposed to parasites over the past year.

A blood sample may be drawn from some participants, depending on whether they have a reaction to the second skin test and whether they have developed skin lesions. The sample is drawn only from patients 18-65 years of age.

Some blood drawn for the study may be used for genetic tests.

DETAILED DESCRIPTION:
The overarching aim of the research program is to develop a vaccine against cutaneous leishmaniasis (CL) based on sandfly salivary proteins (SFSPs). In order to determine whether vaccination with SFSPs can reduce the subsequent incidence of Leishmania major infections or CL in humans, it is first necessary to establish baseline rates of parasite infection and disease. We have selected two rural villages in central Mali where we have readily observed CL lesions in individuals of all ages and large numbers of sandflies that are known to transmit L. major in West Africa. The main objectives of this study are to estimate a cross-sectional prevalence of L. major exposure; to determine the prevalence of CL; to determine an annual incidence rate of L. major infection; and to determine whether robust in vitro T and B cell responses to SFSPs correlate with protection against newly acquired L. major infection or CL. To meet these objectives, a standard leishmanin skin test (LST) will be administered to all residents of two Malian villages in order to identify a cohort of subjects who are at risk for newly acquired L. major. After the sandfly biting and disease transmission seasons, all subjects will be examined for the development of CL lesions every month for 5 months total. CL lesions will be treated topically with paromomycin- methylbenzethonium chloride ointment twice daily for 20 days. Response to therapy will be documented on days 28 and 42 of the protocol. After allowing adequate time for the development of delayed-type hypersensitivity responses to parasite antigens, LSTs will be re-administered to all subjects. Conversion from a negative to positive LST will be taken as evidence of newly acquired L. major infection. LST conversion data and clinical diagnosis of CL lesions will allow us to calculate both the incidence of new L. major infections and CL in our study population. In vitro T and B cell responses to SFSPs will be measured from a subset of individuals and correlated with relative resistance to both L. major infection and the development of clinically apparent lesions.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Only consented volunteers who are permanent residents of Kemena or Sougoula, and who do not have known sensitivity to thiomerosal, will be invited to participate in this study. Otherwise, inclusion criteria specific for each phase of this study are as follows:

Administration of LST, April-May 2006:

Age greater than or equal to 1

Active and passive detection of CL, August-December 2006:

LST negative status in April 2006.

Aspiration of CL lesions, August-December 2006:

Age greater than or equal to18 years, AND

Presence of one or more clinically diagnosed CL lesion

Re-administration of LST in February-March 2007:

LST negative status in April 2006

Collection of whole blood for immunological studies, May 2007 - May 2008:

Age greater than or equal to 3 years and less than or equal to 65 years, AND

LST negative status in February-March 2007.

Active detection of CL, May 2007- May 2008:

LST negative status in February-March 2007.

Aspiration of CL lesions, May 2007 - May 2008:

Age greater than or equal to 3 years, AND

Presence of at least one PCR-diagnosed CL lesion.

Collection of fingerprick blood sample, January-March 2008:

Currently or previously enrolled on protocol

Re-administration of LST, June-July 2008:

LST negative status in February-March 2007.

Collection of whole blood for immunological studies, June - August 2008:

Age greater than or equal to 3 years and less than or equal to 65 years, AND

LST negative status in February-March 2007, AND

One of the following:

Conversion from negative to positive LST reaction during the study period, OR

Occurrence of greater than or equal to 1 PCR-confirmed CL lesion during 10-month survey period, regardless of June-July 2008 LST result, OR

Repeat LST negative result and absence of PCR-confirmed CL lesion during 10-month surveillance period.

Collection of whole blood from healthy volunteers naturally exposed to P. duboscqi October 2008-October 2012

Aqe greater than or equal to 11 years and less than or equal to 65 years, AND resident of Kemena or Sougoula OR patient with a Giemsa stain-confirmed CL lesion beinq evaluated and treated bY study physicians at CNAM in Bamako.

Exposure of individuals to the bites of laboratory-reared, noninfected P. duboscai October 2008-October 2012

Age greater than or equal to 1 years and less than or equal to 65 years AND resident of Kemena or Souaoula.

Dermal biopsy of DTH reactions occurring in individuals exposed to the bites of laboratory-reared, noninfected P. duboscai October 2008- October 2012

Age 18-65 years AND resident of Kemena or Souqoula.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1593 (Actual)
Dates: Start 2006-03-16; Study Completion 2012-09-17

CONTACTS AND LOCATIONS:
Overall Officials: Rick M Fairhurst, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Faculty of Medicine Pharmacy and Dentistry, Bamako, Mali

REFERENCES:
- [Background] Herwaldt BL. Leishmaniasis. Lancet. 1999 Oct 2;354(9185):1191-9. doi: 10.1016/S0140-6736(98)10178-2. PMID 10513726
- [Background] Mahe A, Cisse IAh, Faye O, N'Diaye HT, Niamba P. Skin diseases in Bamako (Mali). Int J Dermatol. 1998 Sep;37(9):673-6. doi: 10.1046/j.1365-4362.1998.00454.x. PMID 9762817
- [Background] el-On J, Halevy S, Grunwald MH, Weinrauch L. Topical treatment of Old World cutaneous leishmaniasis caused by Leishmania major: a double-blind control study. J Am Acad Dermatol. 1992 Aug;27(2 Pt 1):227-31. doi: 10.1016/0190-9622(92)70175-f. PMID 1430361
- [Derived] Coulibaly CA, Traore B, Dicko A, Samake S, Sissoko I, Anderson JM, Valenzuela J, Traore SF, Faye O, Kamhawi S, Oliveira F, Doumbia S. Impact of insecticide-treated bednets and indoor residual spraying in controlling populations of Phlebotomus duboscqi, the vector of Leishmania major in Central Mali. Parasit Vectors. 2018 Jun 14;11(1):345. doi: 10.1186/s13071-018-2909-2. PMID 29898753
- [Derived] Oliveira F, Doumbia S, Anderson JM, Faye O, Diarra SS, Traore P, Cisse M, Camara G, Tall K, Coulibaly CA, Samake S, Sissoko I, Traore B, Diallo D, Keita S, Fairhurst RM, Valenzuela JG, Kamhawi S. Discrepant prevalence and incidence of Leishmania infection between two neighboring villages in Central Mali based on Leishmanin skin test surveys. PLoS Negl Trop Dis. 2009 Dec 15;3(12):e565. doi: 10.1371/journal.pntd.0000565. PMID 20016847